CLINICAL TRIAL: NCT00474708
Title: The Efficacy of Venlafaxine XR (Efexor XR®) Versus SSRIs & Conventional Antidepressants in Depressed Patients Switched From Prior Antidepressants in Psychiatric Outpatient Care Settings in China
Brief Title: Study Comparing the Efficacy of Venlafaxine XR Vs. SSRIs and Conventional Antidepressants in Depressed Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0600B2-4418
Record Dates: First submitted 2007-05-10; First posted 2007-05-17 (Estimated); Results first posted 2010-04-30 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 1.Effexor XR Group
  Interventions: Drug: Effexor
- 2 (Active Comparator): 2.SSRI or Conventional Antidepressant Group
  Interventions: Drug: SSRI

INTERVENTIONS:
Drug: Effexor
  Arms: 1
Drug: SSRI
  Arms: 2

SUMMARY:
This study is an open-label, randomized, multi-center study conducted in a typical psychiatric outpatient practice in China. This study is intended to collect data on the efficacy and safety of venlafaxine XR (Efexor XR®) versus SSRIs and conventional antidepressants in depressed patients that previously failed antidepressant treatment. This data will be used to guide psychiatrists on recommendations for clinic use.

ELIGIBILITY:
Main Inclusion Criteria:

* Males or females, 18 -65 years of age
* Outpatients
* Major depressive disorder based on DSM-IV criteria
* The baseline score of 17-item HAM-D³17
* Switchers from prior antidepressants, who have had no satisfactory improvement (normally after a minimum of 8weeks of treatment), with an approved antidepressant medication or have experienced intolerance due to side effects to their antidepressant medication based on clinical discretion
* Provide written informed consent
* If female is of childbearing potential, must be confirmed no pregnancy at baseline, and use a medically acceptable method of contraception throughout the study.

Main Exclusion Criteria:

* Hypersensitivity to venlafaxine;
* Clinically significant renal or hepatic disease or any other medical disease that, in the opinion of the investigator, might compromise the study, including seizure
* Alcohol or drug abuse within the last year
* A recent history of myocardial infarction or unstable heart disease (within 6 months of baseline)
* Bipolar disorder
* For female, known or suspected pregnancy or breast feeding
* Use of a monoamine oxidase inhibitor (MAOI) within 14 days of baseline; use of any investigational drug within 30 days of baseline.
* Patients have prior use of venlafaxine or use of venlafaxine for the current episode.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1151 (Actual)
Dates: Start 2007-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (14):
- China (14):
  - Beijing, Beijing Municipality
  - Guangzhou, Guangdong
  - Zhengzhou, Henan
  - Wuhan, Hubei
  - Changsha, Hunan
  - Nanjing, Jiangsu
  - Shenyang, Liaoning
  - Jinan, Shandong
  - Shanghai, Shanghai Municipality
  - Xian, Shanxi
  - Tianjin, Tianjin Municipality
  - Hangzhou, Zhejiang
  - Huzhou, Zhejiang
  - Suzhou, Zhejiang

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in China from March 2007 to January 2008.
Pre-assignment Details: There was no screening period for this study. Screening was done by the investigator.
Groups:
- Venlafaxine XR: 75-225 mg per day
- SSRI or Conventional Antidepressant Group: Selective serotonin reuptake inhibitor (SSRI) or Conventional Antidepressants, dependent upon the selected antidepressant, dosages ranging from 20 mg to 250 mg.
Period: Overall Study
Arm/Group | Venlafaxine XR | SSRI or Conventional Antidepressant Group
Started | 791 | 367
Completed | 734 | 342
Not Completed | 57 | 25
Not completed — Lack of Efficacy | 11 | 5
Not completed — Suicide ideation/behavior | 0 | 1
Not completed — Withdrawal by Subject | 7 | 0
Not completed — Lack of compliance | 12 | 4
Not completed — Lost to Follow-up | 18 | 9
Not completed — Physician Decision | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Venlafaxine XR | SSRI or Conventional Antidepressant Group | Total
Number analyzed (Participants) | 787 | 364 | 1151
Age Continuous [Mean (Standard Deviation); unit: years] | 39.97 (12.84) | 40.49 (13.08) | 40.13 (12.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 460 | 225 | 685.0
  Male | 327 | 139 | 466.0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving Remission
Description: Remission is defined as a Hamilton Psychiatric Rating Scale for Depression (HAM-D17) score of ≤ 7. HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Individual items are scored on a 0 to 2 or 4 scale (0=none/absent and 4=most sever) for a maximum total score of 50.
Time Frame: 12 weeks
Population: The analysis population is the per protocol population, consisting of patients who have received at least one dose and have completed the 12 week clinical assessment.
Measure: Number; unit: participants
Arm/Group | Venlafaxine XR | SSRI or Conventional Antidepressant Group
Number analyzed (Participants) | 664 | 295
participants | 554 | 207

2. Secondary Outcome: Number of Patients Achieving Remission (by Co-morbid Anxiety Disorder Status)
Description: as for outcome 1
Time Frame: 12 weeks
Population: The analysis population is the per protocol population, consisting of patients who have received at least one dose and have completed the 12 week clinical assessment. A total of 125 (VEN XR=83, SSRI=42) patients had a co-morbid anxiety disorder and 834 (VEN XR=581, SSRI=253) did not.
Measure: Number; unit: participants
Arm/Group | Venlafaxine XR | SSRI or Conventional Antidepressant Group
Number analyzed (Participants) | 664 | 295
participants
  Co-morbid anxiety disorder | 60 | 23
  No anxiety disorder | 494 | 184

ADVERSE EVENTS:
Arm/Group | Venlafaxine XR | SSRI or Conventional Antidepressant Group
Serious Adverse Events (participants affected / at risk) | 3 | 1
Other Adverse Events (participants affected / at risk) | 418 | 236
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Venlafaxine XR | SSRI or Conventional Antidepressant Group
Attempted suicide (Psychiatric disorders) | 1/787 | 0/365
Pregnancy (Reproductive system and breast disorders) | 1/787 | 0/365
Hospitalization (Psychiatric disorders) | 1/787 | 1/365
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Venlafaxine XR | SSRI or Conventional Antidepressant Group
Constipation (Gastrointestinal disorders) | 66/787 | 43/365
Irritable bowel syndrome (Gastrointestinal disorders) | 1/787 | 0/365
Nausea (Gastrointestinal disorders) | 65/787 | 47/365
Diarrhea (Gastrointestinal disorders) | 7/787 | 6/365
Dry mouth (Gastrointestinal disorders) | 48/787 | 24/365
Bitter taste (Gastrointestinal disorders) | 3/787 | 0/365
No appetite (Gastrointestinal disorders) | 2/787 | 4/365
Vomiting (Gastrointestinal disorders) | 8/787 | 2/365
Stomach disorder (Gastrointestinal disorders) | 4/787 | 1/365
Gastrointestinal disorder (Gastrointestinal disorders) | 2/787 | 6/365
Gastrointestinal reaction (Gastrointestinal disorders) | 3/787 | 0/365
Flatulence (Gastrointestinal disorders) | 7/787 | 7/365
Stomach ache (Gastrointestinal disorders) | 0/787 | 1/365
Dyspepsia (Gastrointestinal disorders) | 2/787 | 0/365
Anorexia (Gastrointestinal disorders) | 4/787 | 5/365
Anesthesia local (Nervous system disorders) | 1/787 | 0/365
Dizziness (Nervous system disorders) | 40/787 | 13/365
Vertigo (Nervous system disorders) | 2/787 | 0/365
Tremor (Nervous system disorders) | 2/787 | 1/365
Night sweats (Nervous system disorders) | 3/787 | 0/365
Sweating increased (Nervous system disorders) | 10/787 | 7/365
Sluggish (Psychiatric disorders) | 1/787 | 0/365
Dreaminess (Psychiatric disorders) | 1/787 | 0/365
Fidget (Psychiatric disorders) | 1/787 | 1/365
Anxiety (Psychiatric disorders) | 2/787 | 7/365
Insomina (Psychiatric disorders) | 7/787 | 8/365
Somnolence (Psychiatric disorders) | 6/787 | 3/365
Sleep disorder (Psychiatric disorders) | 0/787 | 1/365
Sexual dysfunction (Psychiatric disorders) | 1/787 | 2/365
Sexual hypoesthesia (Psychiatric disorders) | 2/787 | 7/365
Drug abuse (Psychiatric disorders) | 1/787 | 0/365
Irritability (Psychiatric disorders) | 1/787 | 0/365
Manic (Psychiatric disorders) | 1/787 | 0/365
Switching (Psychiatric disorders) | 1/787 | 2/365
Suicide (Psychiatric disorders) | 1/787 | 0/365
Dreaming abnormal (Psychiatric disorders) | 1/787 | 0/365
Fever (General disorders) | 1/787 | 0/365
Feeble (General disorders) | 7/787 | 1/365
Abdominal disorder (General disorders) | 1/787 | 0/365
Muscular soreness (General disorders) | 0/787 | 1/365
Fatigue (General disorders) | 10/787 | 3/365
General malaise (General disorders) | 1/787 | 0/365
Head malaise (General disorders) | 2/787 | 0/365
Headache (General disorders) | 21/787 | 0/365
Chest pain (General disorders) | 1/787 | 0/365
Waist disorder (General disorders) | 1/787 | 0/365
Hypertension (Cardiac disorders) | 3/787 | 1/365
Tachycardia (Cardiac disorders) | 0/787 | 1/365
Palpitations (Cardiac disorders) | 12/787 | 5/365
Unstable blood pressure (Cardiac disorders) | 1/787 | 0/365
Hyperlipaemia (Metabolism and nutrition disorders) | 4/787 | 2/365
Thirst (Metabolism and nutrition disorders) | 0/787 | 1/365
Weight increase (Metabolism and nutrition disorders) | 1/787 | 6/365
Weight decrease (Metabolism and nutrition disorders) | 5/787 | 0/365
Leucopenia (Blood and lymphatic system disorders) | 2/787 | 7/365
Hepatic function abnormal (Hepatobiliary disorders) | 4/787 | 4/365
Amenorrhoea (Reproductive system and breast disorders) | 4/787 | 0/365
Pregnancy (Reproductive system and breast disorders) | 1/787 | 0/365
Oligiomenorrhea (Reproductive system and breast disorders) | 2/787 | 0/365
Menstrual disorder (Reproductive system and breast disorders) | 1/787 | 0/365
Micturition frequency (Renal and urinary disorders) | 3/787 | 0/365
Dysuria (Renal and urinary disorders) | 2/787 | 1/365
Micturition disorder (Renal and urinary disorders) | 1/787 | 0/365
Visual abnormal (Eye disorders) | 3/787 | 0/365
Eye disorder (Eye disorders) | 2/787 | 0/365
Dry eye (Eye disorders) | 2/787 | 0/365
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/787 | 2/365
Muscel spasm (Musculoskeletal and connective tissue disorders) | 1/787 | 0/365
Waist pain (Musculoskeletal and connective tissue disorders) | 2/787 | 0/365
Pruritus (Skin and subcutaneous tissue disorders) | 4/787 | 0/365
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3/787 | 0/365
Ejaculation disorder (Reproductive system and breast disorders) | 2/787 | 1/365
Tinnitus (Ear and labyrinth disorders) | 1/787 | 2/365

LIMITATIONS AND CAVEATS:
365 participants were assessed for safety. Certain demographic data (gender and age) is missing for one participant. Thereby resulting in the participant flow reflecting 364 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.